CLINICAL TRIAL: NCT04405700
Title: Measuring Adverse Pregnancy and Newborn Congenital Outcomes: An IeDEA Collaboration Study
Brief Title: Measuring Adverse Pregnancy and Newborn Congenital Outcomes
Acronym: MANGO
Status: Recruiting | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, John Moore Humphrey, Assistant Professor of Medicine, Indiana University
Other Study IDs: 2002126816
Record Dates: First submitted 2020-05-22; First posted 2020-05-28 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: HIV/AIDS; Pregnancy Related; Congenital Disorders; Newborn Morbidity
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Congenital, Hereditary, and Neonatal Diseases and Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort 1 (C1): Prospective recruitment of pregnant women enrolling in antenatal clinic (ANC) at the site. All HIV+ pregnant women and a 1:1 systematic sample of HIV- pregnant women enrolling in ANC at the site will be prospectively enrolled. In addition, medical record data for the mother and infant will be collected at the time of delivery for all women who deliver at the site and as such will contribute to a subset of C2 (below). Women enrolled in C1 who do not deliver at the site will be contacted by phone and through field follow-up to ascertain their pregnancy and infant outcomes. Infants born to women enrolled in this component who are suspected of having congenital abnormalities (CAs) will be enrolled as outlined in C3 (below) if their mothers deliver at the site. If their mothers do not deliver at the site these infants will be enrolled in the field. Photos/videos of infants with CAs will also be taken for review and classification by a panel of experts (see C3 below).
  Interventions: Other: Pharmacovigilance surveillance program
- Cohort 2 (C2): Cross-sectional data collection for deliveries at the site. Data will be collected retrospectively from medical records for all women who deliver at the site (including the women enrolled in C1 above), as well from the medical records of all newborn infants and stillbirths delivered at the site. Missing or incomplete information in the woman or her infant's medical record will be clarified by contacting the woman to provide this information.
  Interventions: Other: Pharmacovigilance surveillance program
- Cohort 3 (C3): Photos/videos of infants with CAs. All newborn infants and stillbirths ≥ 24 weeks gestational age delivered at the site, as well as all infants born to women enrolled in C1, will be assessed by surface exam for the presence of CAs. Video and photographs will be taken of CAs identified on surface exam. These images will be reviewed and classified by panel of experts in genetics, dysmorphology and teratology. Mothers of infants with major CAs will be contacted by phone at 1, 6, and 12 months post-delivery to ascertain their infants' vital status and care engagement status.
  Interventions: Other: Pharmacovigilance surveillance program

INTERVENTIONS:
Other: Pharmacovigilance surveillance program — The pharmacovigilance (PV) surveillance program will prospectively monitor for adverse pregnancy and infant outcomes, including the presence of congenital abnormalities, among HIV-positive and HIV-negative women and their infants at clinical sites affiliated with the International Epidemiology Databases to Evaluate consortium (IeDEA).

SUMMARY:
The purpose of this study is to develop a pharmacovigilance (PV) surveillance program to monitor adverse pregnancy and infant outcomes, including the presence of congenital abnormalities, among HIV-positive and HIV-negative women and their infants at clinical sites affiliated with the International Epidemiology Databases to Evaluate consortium (IeDEA).

DETAILED DESCRIPTION:
In part 1 of this study, the investigators will use a mixed prospective and cross-sectional cohort study design to implement a PV program at two health facilities affiliated with the Academic Model Providing Access to Healthcare (AMPATH) in western Kenya. The investigators will analyze these data to examine any associations between antiretroviral treatment (ART) and (a) pregnancy and (b) infant/birth outcomes. In part 2, the investigators will create standardized protocols and data exchange standards within IeDEA to enable the merging and analysis of multiregional IeDEA PV data. This will include establishing a Data Coordinating Center based at Indiana University (IU) to serve as a hub for collecting, disseminating and archiving data from the study in Kenya as well as data collected through a similar, ongoing study at health facilities in South Africa affiliated with IeDEA. This study will establish a multiregional PV infrastructure within IeDEA that can be further scaled within the broader IeDEA network.

ELIGIBILITY:
C1. Prospective recruitment of HIV+ and HIV- pregnant women enrolling in ANC at the site:

Inclusion criteria for women

1. Pregnant and enrolled in ANC at the study site;
2. Understands English or Swahili.

Exclusion criteria for women a. Any physical or mental disability that prevents the woman from providing informed consent

Inclusion criteria for infants

a. All infants at any gestational age who are born to enrolled women will be included Exclusion criteria for infants (none)

C2. Data collection for all deliveries at the site:

Inclusion criteria for women a. Woman delivers at the site and the delivery is registered at the site

Exclusion criteria for women (none)

Inclusion criteria for live/stillborn infants

a. Infant is delivered at the site and results in the infant/stillbirth being registered at the site

Exclusion criteria for infants (none)

C3. Photos/videos of infants with CAs:

Inclusion criteria for infants

1. The infant is live or stillborn at ≥ 24 weeks estimated gestational age
2. The infant has a suspected CA on surface exam

Exclusion criteria for infants (none)

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant and postpartum women who are HIV+ and HIV- and their infants.
Sampling Method: Probability Sample
Enrollment: 2800 (Estimated)
Dates: Start 2020-09-29 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Pregnancy outcomes | At time of delivery
  Live Birth, Still Birth, Miscarriage, Termination of pregnancy, Ectopic Pregnancy, Molar Pregnancy, Not Pregnant, Other); also including pre-term delivery (<37 weeks gestational age) or very pre-term delivery (<32 weeks gestational age)
Infant/birth outcomes | At 1, 6, and 12 months post-delivery
  Congenital abnormalities on newborn surface exam (e.g., extra digit, hydrocephalus, skull defects, eyes, face, mouth/lip/palate, chest, abdomen, anus, limbs, spine (including neural tube defects), hips, genitalia, skin, etc.); also including low birth weight, small for gestational age (<10th percentile) or very small for gestational age (<3rd percentile)

CONTACTS AND LOCATIONS:
Locations (1):
- Moi Teaching and Referral Hospital, Eldoret, Kenya

IPD SHARING:
Plan to Share IPD: No